CLINICAL TRIAL: NCT03451604
Title: Time Involved in Patient Information During Preoperative Assessment Clinic and Ratio Between Evaluation and Information Times
Brief Title: PAC Time Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Principal Investigator, Vincent COMPERE, professor, University Hospital, Rouen
Other Study IDs: E2016-74
Record Dates: First submitted 2018-01-02; First posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Anesthesia; Assessment Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: preoperative assessement — All data concerning study, involved in normal care of patient for his anesthesia (non interventional study), where included in anonymous computerized database by anesthesiologist during pre operative clinic.

SUMMARY:
The aim of the preoperative assessment clinic (PAC) is to ensure optimal anaesthesia, reduce the morbidity associated with surgery, to increase the quality and decrease the cost of perioperative care 1. In addition, the PAC is an appropriate time to educate the patient on anaesthesia, perioperative care, and pain treatments, to reduce anxiety, to develop care plans, and to obtain informed consent. Moreover, a strong correlation exists between the time spent at the PAC and patient satisfaction2,3.

A high variability of preoperative assessment clinic (PAC) times is a reason for waiting time for patient. A better match between the reserved PAC time and the real consultation time could improved efficiency in consultation theatre. The PAC time depends on various parameters. On average the preoperative assessment of patients with a higher American Society Anesthesiologists' (ASA) class requires more time 4. In other monocentric study, the mean (SD) procedure time was 13 (6) min for the physician. It was significantly longer for patients with a higher ASA class : 10 min for ASA I, 14 min for ASA II, 17 min for ASA III and 21 min for ASA IV patients. In this monocentric study, every patient had a nurse consultation before PAC by the anesthesiologist.

The primary endpoint of this study was to assess the time involved in preoperative assessment clinic included the time during patient's health status has to be assessed (this encompasses a medical history and physical examination) and the time during the patient education on anaesthesia, perioperative care and pain treatments, to reduce anxiety, to develop care plans and to obtain informed consent.

ELIGIBILITY:
Inclusion Criteria:

- Patients scheduled to undergo elective surgery under general or regional anaesthesia

Exclusion Criteria

* patients under 16 years of age
* emergency surgery

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients scheduled to undergo elective surgery under general or regional anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
total time involved in preoperative anesthesia consultation (min) | 30 min
  total time (min) is defined by the time between patient entry and discharge from the consultation office. It integrates time for patient assessment (this encompasses a medical history and physical examination) and time for patient information on the benefits and risks of the chosen anesthetic strategy (patient education on anaesthesia, perioperative care and pain treatments, to reduce anxiety, to develop care plans and to obtain informed consent)

SECONDARY OUTCOMES:
anesthesia and surgery information and patient demographics | 30 min
  Data included anesthesia and surgery information and patient demographics
  * ASA status
  * Age
  * BMI
  * In patient or outpatient
  * Number of medication
  * Number of co morbidity
  * Socioeconomic level
  * Surgical specialty
  * Senior or resident anesthesiologist (year experience)
  * Preoperative anxiety between 0 and 10
  * Patient satisfaction between 0 and 10

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No